CLINICAL TRIAL: NCT03958851
Title: Measurement of Renal Artery Resistive Index as a Predictor of Severity of Lupus Nephritis and Its Response to Treatment
Brief Title: Renal Resistive Index as a Marker of Severity and Treatment Outcomes in Lupus Nephritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasser Abd Elmawgood Fysal Ibrahim, assistant lecturer, Assiut University
Other Study IDs: RRI in lupus nephritis
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Lupus Nephritis
Keywords: renal resistive index
MeSH Terms: conditions — Lupus Nephritis | interventions — Kidney Function Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with lupus nephritis: Lupus nephritis is diagnosed by either the presence of proteinuria (>0.5 g/day), active urinary sediment (with red blood cell, granular, tubular and/or mixed casts), or an unexplained rise in serum creatinine in patients with systemic lupus.
  Interventions: Diagnostic Test: Doppler ultrasonography of renal arteries; Diagnostic Test: Renal biopsy; Diagnostic Test: kidney function tests; Diagnostic Test: The 24-hour urine protein test; Diagnostic Test: complete blood counting (CBC)
- systemic lupus patients without lupus nephritis: The diagnosis of SLE will be according to the 1997 American college of Romatology revised criteria (Hochberg 1997).these group will be taken as a control group
  Interventions: Diagnostic Test: Doppler ultrasonography of renal arteries
- healthy individuals: a group of age and sex matched healthy individuals will be taken as a control group.
  Interventions: Diagnostic Test: Doppler ultrasonography of renal arteries

INTERVENTIONS:
Diagnostic Test: Doppler ultrasonography of renal arteries — Ultrasound evaluation will be performed for all patients as well as healthy individuals.in patients with lupus nephritis,the ultrasound evaluation will be performed the 24 h prior to the renal biopsy . In the maximum long-axis section images, the largest diameter and width of each kidney will be measured. The participants will be scanned in a supine or decubitus position to achieve an ultrasound beam as close to parallel to the blood flow direction in the intrarenal artery as possible. RRI is measured as :
  RRI = (peak systolic velocity - end diastolic velocity ) / peak systolic velocity. the average of three measurements will be taken.
Diagnostic Test: Renal biopsy — Renal biopsy is a medical procedure in which a small piece of kidney is removed from the body for examination, usually under a microscope. Microscopic examination of the tissue can provide information needed to diagnose, monitor or treat problems of the kidney.Renal biopsy will be taken according American college of Romatology guidelines 2012.The renal biopsy samples were evaluated according to the Revision of the International Society of Nephrology/Renal Pathology Society classification for lupus nephritis 2017. the actvity index and chronicity index will be calculated.
  Groups: patients with lupus nephritis
Diagnostic Test: kidney function tests — blood sample will be taken to measure blood urea nitrogen (BUN) and serum creatinine(S Cr). estimated glomerular filtration rate (eGFR) will be measured using CKD-EPI Equation.These investigations will be done at the beginning of the study and every month for sex months for each patient to determine degree of response to treatment .
  Groups: patients with lupus nephritis
Diagnostic Test: The 24-hour urine protein test — The 24-hour urine protein test checks how much protein is being spilled into the urine.Urine samples are collected in one or more containers over a period of 24 hours. The containers are kept in a cool environment and then sent to a lab for analysis. Specialists then check the urine for protein.This investigations will be done at the beginning of the study and every month for sex months for each patient to determine degree of response to treatment .
  Groups: patients with lupus nephritis
Diagnostic Test: complete blood counting (CBC) — A complete blood count is a blood panel that gives information about the cells in a patient's blood, such as the cell count for each blood cell type and the concentrations of hemoglobin.
  Groups: patients with lupus nephritis

SUMMARY:
All patients with SLE that will be admitted in internal medicine department from August 2019 to January 2021 are eligible to be targeted and included in the study. The diagnosis of SLE will be according to the 1997 American college of Romatology revised criteria (Hochberg 1997). SLE patients with lupus nephritis will take kidney biopsy for standard care of management according to American college of Romatology guidelines 2012. The study will include three groups as follow:

1 - SLE patients with lupus nephritis. 2- SLE patients without lupus nephritis 3-A group of age and sex matched healthy individuals. The first group will represent the study group while the second and third groups group will be taken as control group Exclusion criteria: patients with

1- Chronic renal failure 2- Diabetes mellitus (DM) 3-Obstructive nephropathy 4- Renal artery stenosis 5- Hypertension 6- Heart failure 7- Hepatic diseases. 8- Existing intra renal A-V fistula. 9-Renal vein thrombosis

Aims of the Research :

1. Assessment of the renal resistive index in patients with lupus nephritis (LN), in SLE patients without lupus nephritis and in the healthy controls.
2. Comparing the renal resistive index values in SLE patients with lupus nephritis with the SLE patients without LN and healthy controls.
3. Assessment of the correlation between renal resistive index (RRI) and histological findings in renal biopsy in patients with lupus nephritis.
4. Assessment of the correlation between renal resistive index (RRI) and renal function parameters (BUN, S Cr and eGFR).
5. Evaluation of the role of RRI as predictor of treatment outcomes in patients with lupus nephritis.

The study will be enrolled in three steps:

The first step:comparison of renal artery resistive index(RRI) values between study group and controls.

The second step :correlation between RRI of the patients with lupus nephritis and histological findings in renal biopsy and/ or kidney function parameters (BUN ,SCr , eGFR).

The third step:the patients with lupus nephritis will be followed up for six month receiving the usual treatment according to KDIGO guidelines 2012 to demonstrate the response to treatment in patient with pathological RRI compared to with normal RRI

DETAILED DESCRIPTION:
LN is known to be one of the most serious complications of SLE and it is the major predictor of poor prognosis. In the United States, approximately 35% of adults with SLE have clinical evidence of nephritis at the time of diagnosis; with an estimated total of 50 to 60% developing nephritis during the first 10 years of disease. Lupus nephritis is diagnosed by either the presence of proteinuria (>0.5 g/day), active urinary sediment (with red blood cell, granular, tubular and/or mixed casts), or an unexplained rise in serum creatinine (S Cr). A kidney biopsy is the gold standard to diagnose LN as it provides information regarding the pattern and severity of renal involvement as well as the stage, activity and chronicity. These are all important considerations influencing treatment decisions. However, the invasive nature make it contraindicated in certain situation like bleeding tendency. In one report, five of seven patients with significant bleeding after renal biopsy were patients with LN. Serial biopsy may be needed to monitor progression and treatment. This will increase risk of complication and may be not practical.

The renal arterial resistive index (RRI) is a sonographic index to assess for renal arterial disease. It is measured as:

RRI = (peak systolic velocity - end diastolic velocity) / peak systolic velocity .The RRI was introduced in 1950, and was initially proposed for the semi-quantitative assay of intra-renal vascular resistance by Gosling and Pourcelot in 1974. RRI is and markedly affected by renal determinants such as renal interstitial and venous pressure. In humans in vivo, the acute increase of renal interstitial pressure by hydronephrosis or of venous pressure by venous thrombosis, or of both by abdominal hypertension, results in a linearly related increase in RRI. Increases in the RRI have been observed in a number of pathological conditions, which increase renal interstitial and venous pressure such as renal allograft acute rejection, parenchymal nephropathies, acute kidney injury, renal artery stenosis, chronic kidney disease (CKD), diabetic nephropathy, obstructive nephropathy. Remarkably, interstitial ﬁbrosis closely correlates to renal function and long term prognosis, and may underlie the role of RRI as an independent marker of renal and clinical outcome in chronic renal diseases. No standard, validated, cut-off to distinguish normal from high RRI has been identified to date. RRI values between 0.7 and 0.85 have been associated with renal functional impairment in patients with chronic kidney disease and stenosis of the renal artery. Previous data have revealed a significant correlation between the increased RRI value (RRI>0.7) and renal functional parameters (creatinine and blood urea nitrogen levels) and/or histological finding, such as glomerulosclerosis, tubulointerstitial damage and vascular lesions. Few studies evaluate the role of RRI as marker of severity in LN and its potential use as non-invasive marker in the assessment of the outcomes and in treatments response. To date, the usefulness of RRI in monitoring the progression and treatment of LN is controversial.

Type of the study: : observational analytic cross sectional study - cohort study (the part of the study in which the patients of LN are followed for six month receiving the usual treatment according to KDIGO( Kidney Disease: Improving Global Outcomes) guidelines 2012 to demonstrate the response to treatment in patient with pathological RRI compared to with normal RRI) - Study Setting: Assiut University Hospital (internal medicine departments)

All patients with SLE that will be admitted in internal medicine department from August 2019 to January 2021 are eligible to be targeted and included in the study. The diagnosis of SLE will be according to the 1997 American college of Romatology revised criteria (Hochberg 1997). SLE patients with lupus nephritis will take kidney biopsy for standard care of management according to American college of Romatology guidelines 2012. The study will include three groups as follow:

1 - SLE patients with lupus nephritis. 2- SLE patients without lupus nephritis 3-A group of age and sex matched healthy individuals. The first group will represent the study group while the second and third groups group will be taken as control group .

Sample Size technique: total coverage The ratio of controls to study group will be 2:1.

Study methods:

A-The study group will be subjected to:-

1. History taking and complete physical examination.
2. Laboratory testing: complete blood counting (CBC), blood urea nitrogen (BUN), serum creatinine(S Cr), serum albumin( ALB) estimated glomerular filtration rate (eGFR) (using CKD-EPI(Chronic Kidney Disease Epidemiology Collaboration) Equation) and 24 h urinary protein excretion. These investigations will be taken at the beginning of the study and every month for sex months to determine degree of response to treatment according to KDIGO guidelines 2012.
3. Renal biopsy will be taken according American college of Romatology guidelines 2012.

   The renal biopsy samples were evaluated by renal pathologists, according to the Revision of the International Society of Nephrology/Renal Pathology Society classification for lupus nephritis 2017. Briefly, chronicity index will be calculated as follows: glomerulosclerosis (GS) <25% of the glomeruli =1; GS = 26-50% of the glomeruli= 2; GS > 50% of the glomeruli =3. Fibrous crescents: Fibrous crescents in <25%of the glomeruli=1, Fibrous crescents in 25-50% of the glomeruli =2, Fibrous crescents in >50% of the glomeruli =3. Tubular atrophy: tubular atrophy in <25% of the cortical tubules=1, tubular atrophy in 25-50% of the cortical tubules 2, tubular atrophy in >50% of the cortical tubules =3. Interstitial fibrosis: interstitial fibrosis in <25% of the cortex=1, interstitial fibrosis in 25-50% of the cortex 2, interstitial fibrosis in >50% of the cortex =3. The chronicity index score range from 0 to 12.

   Activity index will be calculated as follow Endocapillary hypercellularity: Endocapillary hypercellularity in <25% of glomeruli =1, 25%-50% of glomeruli =2, or >50% of glomeruli =3. Neutrophils/karyorrhexis : Neutrophils and/or karyorrhexis in <25% of glomeruli =1*2, 25%-50% of glomeruli =2*2 or >50 of glomeruli =3 *2.Fibrinoid necrosis : Fibrinoid necrosis in <25% of glomeruli =1*2,25%-50% of glomeruli =2*2 or >50% of glomeruli =3*2.Hyaline deposits: Wire loop lesions and/or hyaline thrombi in <25% of glomeruli =1,25%-50% of glomeruli =2 or >50% of glomeruli = 3. Cellular/ﬁbrocellular crescents: Cellular and/or ﬁbrocellular crescents in <25% of glomeruli=1, 25%-50% of glomeruli =2 or >50% of glomeruli =3. Activity index score range from 0 to 24.
4. Doppler ultrasonography. Ultrasound evaluation will be performed 24 h prior to the renal biopsy for all patients and healthy individuals. In the maximum long-axis section images, the largest diameter and width of each kidney will be measured. The participants will be scanned in a supine or decubitus position to achieve an ultrasound beam as close to parallel to the blood flow direction in the intrarenal artery as possible. An ultrasound probe covered with transmission gel will be gently placed on the skin over the kidneys. The PSV, EDV and RI will be measured.

B-The control group (non renal SLE patients and healthy individuals) will be subjected to history taking, physical examination and Doppler ultrasonography as the same as the study group.

Aims of the work:

1. Assessment of the renal resistive index in patients with lupus nephritis (LN), in SLE patients without lupus nephritis and in the healthy controls.
2. Comparing the renal resistive index values in SLE patients with lupus nephritis with the SLE patients without LN and healthy controls.
3. Assessment of the correlation between renal resistive index (RRI) and histological findings in renal biopsy in patients with lupus nephritis.
4. Assessment of the correlation between renal resistive index (RRI) and renal function parameters (BUN, S Cr and eGFR).
5. Evaluation of the role of RRI as predictor of treatment outcomes in patients with lupus nephritis.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with lupus nephritis that will be admitted in internal medicine department from August 2019 to January 2021 .
2. All patients with systemic lupus erythematosus(SLE) without renal affection, that will be admitted in internal medicine department from August 2019 to January 2021 .
3. A group of age and sex matched healthy individuals. The first group is the study group while the second and third groups group will be taken as control group

Exclusion Criteria:

1. chronic renal failure
2. Diabetes mellitus
3. Obstructive nephropathy
4. Renal artery stenosis
5. Hypertension
6. Heart failure
7. Hepatic diseases.
8. Existing intra renal A-V fistula.
9. Renal vein thrombosis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients with SLE that will be admitted in internal medicine department from August 2019 to January 2021 are eligible to be targeted and included in the study. The diagnosis of SLE will be according to the 1997 American college of Romatology revised criteria (Hochberg 1997). SLE patients with lupus nephritis will take kidney biopsy for standard care of management according to American college of Romatology guidelines 2012.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
The mean of renal artery resistive(RRI) in each group | 30 minutes
  the sum of RRI values in each group divided by the number of individuals in each group
Correlation between Renal Resistive Index and chronicity index in renal biopsy of patients with Lupus Nephritis | one weak
  Renal Resistive Index will be measured as :RRI = (peak systolic velocity - end diastolic velocity ) / peak systolic velocity .chronicity index score in renal biopsy will be calculated according to the Revision of the International Society of Nephrology/Renal Pathology Society classification for lupus nephritis 2017. Result of renal biopsy will be reported within one weak.Correlation between RRI and chronicity index using correlation tests using SPSS version 20; pearson correlation test if the data are normally distributed and spearman correlation test if the data aren't normally distributed

SECONDARY OUTCOMES:
The mean of renal artery resistive index in each histological class in renal biopsy | one weak
  pathological RRI(RRI>0.7) .Renal biopsy will be evaluated according to the Revision of the International Society of Nephrology/Renal Pathology Society classification for lupus nephritis 2017. There are 6 classes of lupus nephritis in renal biopsy. Number of patients in each class will be identified. the sum of RRI values in each class divided by the number of patients in each class
Correlation between renal artery resistive index (RRI) and renal function parameters (BUN, SCr and eGFR) in patients with lupus nephritis | two hours
  measurement of RRI in each patient with lupus nephritis . Blood sample from the same patient to measure blood urea nitrogen (BUN), serum creatinine(S Cr) and estimated glomerular filtration rate (eGFR) (using CKD-EPI Equation)
Correlation between renal artery resistive index and response to treatment in patients with lupus nephritis | 6months
  RRI will be measured for every patient with lupus nephritis at the beginning of the study. the patients will be followed for 6 months .BUN,S Cr , eGFR and and 24 h urinary protein excretion will be measured at the beginning of the study and every month for sex months to determine degree of response to treatment in patients with pathological RRI(0.7) compared to those with normal RRI.
Correlation between RRI and mean of hemoglobin level in patients with lupus nephritis. | 6 months
  RRI will be measured for every patient of lupus nephritis at the beginning of the study.Hemoglobin level will be measured at the beginning of the study and every month for sex months and the mean will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf A Elshazly, professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boddi M, Natucci F, Ciani E. The internist and the renal resistive index: truths and doubts. Intern Emerg Med. 2015 Dec;10(8):893-905. doi: 10.1007/s11739-015-1289-2. Epub 2015 Sep 4. PMID 26337967
- [Background] Krumme B. Renal Doppler sonography--update in clinical nephrology. Nephron Clin Pract. 2006;103(2):c24-8. doi: 10.1159/000090605. Epub 2006 Mar 10. PMID 16543752
- [Background] Hahn BH, McMahon MA, Wilkinson A, Wallace WD, Daikh DI, Fitzgerald JD, Karpouzas GA, Merrill JT, Wallace DJ, Yazdany J, Ramsey-Goldman R, Singh K, Khalighi M, Choi SI, Gogia M, Kafaja S, Kamgar M, Lau C, Martin WJ, Parikh S, Peng J, Rastogi A, Chen W, Grossman JM; American College of Rheumatology. American College of Rheumatology guidelines for screening, treatment, and management of lupus nephritis. Arthritis Care Res (Hoboken). 2012 Jun;64(6):797-808. doi: 10.1002/acr.21664. No abstract available. PMID 22556106
- [Background] Rees F, Doherty M, Grainge MJ, Lanyon P, Zhang W. The worldwide incidence and prevalence of systemic lupus erythematosus: a systematic review of epidemiological studies. Rheumatology (Oxford). 2017 Nov 1;56(11):1945-1961. doi: 10.1093/rheumatology/kex260. PMID 28968809
- [Result] Chen Q, He F, Feng X, Luo Z, Zhang J, Zhang L, Wang Y, Tong J. Correlation of Doppler parameters with renal pathology: A study of 992 patients. Exp Ther Med. 2014 Feb;7(2):439-442. doi: 10.3892/etm.2013.1442. Epub 2013 Dec 10. PMID 24396421
- [Result] Corapi KM, Dooley MA, Pendergraft WF 3rd. Comparison and evaluation of lupus nephritis response criteria in lupus activity indices and clinical trials. Arthritis Res Ther. 2015 Apr 28;17(1):110. doi: 10.1186/s13075-015-0621-6. PMID 25927414
- [Result] Tao JL, Li H, Li C, Xu XW, Li JF, Yi N, Liu DY, Qin Y, Cai JF, Liu BY, Xu H, Gao RT, Ye WL, Ye W, Li XM, Li XW. [Risk factors of post-renal biopsy bleeding]. Zhongguo Yi Xue Ke Xue Yuan Xue Bao. 2008 Jun;30(3):313-7. Chinese. PMID 18686612
- [Result] Sugiura T, Nakamori A, Wada A, Fukuhara Y. Evaluation of tubulointerstitial injury by Doppler ultrasonography in glomerular diseases. Clin Nephrol. 2004 Feb;61(2):119-26. doi: 10.5414/cnp61119. PMID 14989631